CLINICAL TRIAL: NCT06170996
Title: Internet-Based Behavioural Parent Training Intervention for Children With Attention-Deficit/Hyperactivity Disorder
Brief Title: Internet-Based Behavioural Parent Training Intervention for Children With Attention Deficit/Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Mental Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2023.0912.02
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Attention deficit hyperactivity disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based behavioral parent training (I-BPT+RCC) (Experimental): Internet-based behavioural parent training in a group format in addition to routine clinical care, 8 sessions over 2 months, delivered by a systematically trained and supervised therapist.
  Interventions: Behavioral: Internet-based behavioral parent training (I-BPT)
- Routine clinical care (RCC) (No Intervention): Routine clinical care for 2 months, delivered by experienced child psychiatrists, including medication treatment and examinations, crisis interventions, parent counselling and support.

INTERVENTIONS:
Behavioral: Internet-based behavioral parent training (I-BPT) — Internet-based behavioural parent training in a group format, 8 sessions over 2 months, delivered by a systematically trained and supervised therapist.
  Arms: Internet-based behavioral parent training (I-BPT+RCC)

SUMMARY:
This study aims to investigate the effectiveness of an Internet-based behavioural parent training intervention on children's ADHD symptoms and children's and parents' mental health status.

DETAILED DESCRIPTION:
The study design was a 2-parallel-group experimental longitudinal study. Firstly, the children received a diagnostic interview by an experienced child and adolescent psychiatrist at Wuhan Mental Health Centre for confirmation of inclusion and exclusion criteria. Parents who were eligible for the inclusion criteria and interested in the internet-based behavioural Parent Training (I-BPT) program were recruited. After the assessments of ADHD symptoms and psychiatric comorbidity, participants were randomly assigned in a 1:1 ratio to either the routine clinical care (RCC) group or I-BPT+RCC group using computer-generated randomization numbers. Participants in the I-BPT+RCC group were offered 2 months (8 weeks) of internet-assisted parent training in addition to routine outpatient treatment. The RCC group initially received only routine outpatient treatment, yet, after post-follow-up assessment, they were provided with the same I-BPT intervention for ethical considerations. Both groups were followed up after intervention by electronic questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 1.Meeting the diagnostic criteria for ADHD in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition
* 2.Total IQ greater than 70 as measured by the Wechsler Intelligence Scale for Children, Fourth Edition (WISC-IV)
* 3.Child and their parents consent to the study

Exclusion Criteria:

* 1.Children or parents with severe organic encephalopathy and other severe mental disorders
* 2.Has received or is receiving behavioral treatment (parent training)
* 3.Parents who could not understand or lacking of access to computers and the Internet

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-03-12 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Chinese version of Swan-son Nolan and Pelham, Version IV Scale-parent form (SNAP-IV) | From baseline to 2 months
  This questionnaire consists of two symptom domains: inattention (9 items) and hyperactivity/impulsivity (9 items). Each item of SNAP-IV assigned a score from 0 (never or rarely) to 3 (very often), with a higher score indicating more severe ADHD symptoms.
Weiss Functional Impairment Scale-Parent form (WFIRS-P) | From baseline to 2 months
  This scale consists of 50 items, each with a score ranging from 0 to 3, a higher average score indicates a greater impairment.

SECONDARY OUTCOMES:
Screen for Child Anxiety Related Emotional Disorders (SCARED) | From baseline to 2 months
  This scale encompasses 41 items, each item ranges from 0 to 2, with a higher score indicating more severe anxiety symptoms.
Children's Depression Inventory-Short Form (CDI-S) | From baseline to 2 months
  The CDI-S consists of 10 items, each scored with 0, 1, or 2 points. Depression is rated on a scale of 0 to 15; higher scores indicate more serious symptoms of depression.
The seven-item version of the Generalized Anxiety Disorder (GAD-7) | From baseline to 2 months
  The GAD is a 7-item self-reported questionnaire, with a total score ranging from 0 to 21, and a higher score indicating increased anxiety.
The nine-item version of the Patient Health Questionnaire (PHQ-9) | From baseline to 2 months
  The PHQ-9 scale comprises nine items, assigning scores from 0 (not at all) to 3 (nearly every day). The total score of the PHQ-9 questionnaire ranged from 0 to 27, with a higher score indicating more severe depressive symptoms.
Parenting Stress Index-Short Form (PSI-SF) | From baseline to 2 months
  This scale consists of 15 items, with a total score from 15 to 75. The higher score indicates more higher stress level.
Client Satisfaction Questionnaire adapted to Internet-based interventions (CSQ-I) | posttest: 2 months to pretest
  The CSQ-I consists of 8 items, with a total score of 0 to 32. The higher scores correspond to greater satisfaction of participants.

CONTACTS AND LOCATIONS:
Overall Officials: Tang Jun, Master, Study Director — director in Child and Adolescent Psychological Ward of Wuhan Mental Health Center
Locations (1):
- Wuhan Mental Health Centre, Wuhan, Hubei, China